CLINICAL TRIAL: NCT00000455
Title: Targeted Naltrexone for Early Problem Drinkers
Brief Title: Naltrexone for Early Problem Drinkers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Dr. Henry R. Kranzler, University of Pennsylvania
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NIAAAKRA11062; R01AA011062 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: naltrexone

SUMMARY:
Early problem drinkers are prevalent in the United States. Recent controlled trials have shown that brief interventions in the primary care setting can reduce drinking and alcohol-related problems in patients who lack evidence of alcohol dependence.

Although naltrexone (Revia) has been approved for the treatment of alcohol dependence, few pharmacotherapy studies have been undertaken with early problem drinkers. This study is an 8-week trial of naltrexone versus placebo, combined with coping skills treatment that either focuses on targeted use of medication or serves as background to daily use of the medication. A total of 160 early problem drinkers recruited through screening in primary care medical settings will be randomly assigned to one of four treatment groups. Followup evaluations will be conducted at the end of treatment and again 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Limited to early problem drinkers (i.e., those with no more than mild alcohol dependence).
* Have an average weekly alcohol consumption of greater than or equal to 24 standard drinks for men and 18 standard drinks for women.
* Able to read English at the eighth grade or higher level and show no evidence of significant cognitive impairment.
* Willing to provide a collateral informant for interviews regarding the patient's drinking during the study.
* A woman of child-bearing potential must be non-lactating, practicing a reliable method of birth control, and have a negative pregnancy test prior to initiation of treatment.
* Willing to provide a signed informed consent to participate in the study.

Exclusion Criteria:

* Have a current clinically significant physical disease or abnormality.
* Have a serious psychiatric illness.
* Have a current diagnosis of drug dependence (other than nicotine dependence) or a lifetime diagnosis of opioid dependence.
* A current diagnosis of alcohol dependence that is moderate or greater in severity or a history of alcohol withdrawal, or recurrent use of alcohol to alleviate alcohol withdrawal symptoms.
* Used opioids or other psychoactive medications regularly in the month prior to study enrollment.
* History of hypersensitivity to naltrexone (Revia).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160
Dates: Study Completion 2002-09

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, University of Pennsylvania, Philadelphia, Pennsylvania, United States